CLINICAL TRIAL: NCT04780932
Title: Initial Dual Oral coMbination Therapy Versus Standard-of-care Initial Oral Monotherapy Prior to Balloon Pulmonary Angioplasty in Patients With Inoperable Chronic Thromboembolic Pulmonary hyperTension
Acronym: IMPACT-CTEPH
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Janssen, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APHP201037
Record Dates: First submitted 2021-02-15; First posted 2021-03-04 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Thromboembolic Pulmonary Hypertension; Chronic Disease; Inoperable Disease
MeSH Terms: conditions — Chronic Disease | interventions — macitentan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Arm (Placebo Comparator): Oral Standard-of care riociguat from Day 1 to Week 42 (+/- 1 week). Posology 1mg tid - 2,5 mg tid. Oral Placebo 10 mg/day from Day 8 (+/- 3 days) to Week 42 (+/- 1 week). At week 16, subjects who are still symptomatic (WHO functional II to IV) and have PVR ≥ 240 dyn.sec.cm-5 will be offered additional treatment by BPA.
  Interventions: Drug: Placebo
- Experimental Arm (Experimental): Oral Standard-of care riociguat from Day 1 to Week 42 (+/- 1 week). Posology 1mg tid - 2,5 mg tid. Oral Macitentan 10 mg/day from Day 8 (+/- 3 days) to Week 42 (+/- 1 week). At week 16, subjects who are still symptomatic (WHO functional II to IV) and have PVR ≥ 240 dyn.sec.cm-5 will be offered additional treatment by BPA.
  Interventions: Drug: Macitentan 10mg

INTERVENTIONS:
Drug: Macitentan 10mg — Macitentan 10 mg will be initiated at Day 8 (+/- 3 days) until week 42 (+/- week). The recommended dose is 10 mg once daily by oral administration
  Arms: Experimental Arm
Drug: Placebo — Placebo 10 mg will be initiated at Day 8 (+/- 3 days) until week 42 (+/- week). The recommended dose is 10 mg once daily by oral administration
  Arms: Control Arm

SUMMARY:
Chronic thromboembolic pulmonary hypertension (CTEPH) is characterised by an obstruction of proximal or more distal pulmonary arteries by residual organized thrombi, combined with a variable microscopic pulmonary vasculopathy (microvasculopathy). Besides lifelong anticoagulation, surgical pulmonary endarterectomy is the treatment of choice in subjects with proximal CTEPH affecting large pulmonary arteries. However, around half of CTEPH subjects are not operated, mainly because of distal lesions inaccessible to surgery. International data have reported survival rates of 88, 79, and 70% at 1, 2, and 3 years, respectively, in subjects with inoperable CTEPH, underscoring the need for better treatment strategies. In those subjects, current guidelines recommend medical therapy with or without balloon pulmonary angioplasty (BPA). Currently, only one drug (riociguat), targeting the NO pathway, is approved and reimbursed in Europe. Thus, riociguat monotherapy is considered as the standard-of-care treatment for subjects newly diagnosed with inoperable CTEPH. Recently, macitentan, targeting the endothelin-1 pathway, showed to be also effective in subjects with inoperable CTEPH. However, macitentan is currently not approved for CTEPH in Europe.

BPA has been also reported to improve hemodynamics, symptoms and exercise capacity. However, complications, including mainly vascular injury, may occur during this procedure and it has been shown that the risk of BPA-related complications was strongly related to the level of pre-BPA mean pulmonary artery pressure (mPAP) and pulmonary vascular resistance (PVR). Medical therapy and BPA have in fact complementary effects since they target different lesions. Indeed, BPA targets fibrotic organized thrombi in the segmental arteries down to small pulmonary arteries of 2-5 mm in diameter. Medical therapy, for its part, targets microvasculopathy, similar to that observed in pulmonary arterial hypertension (PAH), in vessels less than 0.5 mm in diameter. Therefore, it is strongly believed that the use of medical therapy prior to BPA may reduce the risk of BPA-related complications by improving pulmonary hemodynamics and may improve global efficacy. In PAH, initial dual oral combination therapy with drugs targeting the NO and endothelin pathways is considered as a standard of care, more efficacious than monotherapy and safe. In contrast, there are no data from controlled trials regarding the efficacy and safety of initial combination therapy regimens versus standard-of-care monotherapy in treatment-naïve subjects with inoperable CTEPH.

The investigators hypothesize that initial dual oral combination therapy may be superior to standard-of-care riociguat monotherapy for improving pulmonary hemodynamics prior to BPA and for reducing the risk of BPA-related complications.

DETAILED DESCRIPTION:
The Screening period will last up 28 days maximum. It begins at the first screening assessment and ends with subject inclusion. The Screening visit date is the date when the first screening assessment is performed.

The Treatment period will start at Day 1 with the first dose of riociguat and ends at Week 42 / End-of-Treatment (EOT) visit.

On Day 8, the experimental treatment with macitentan / placebo will be started.

During this period, regular hospital visits will be performed (Week 16, Week 29).

In addition, laboratory tests will be performed every 4 weeks as part of standard of care.

Subjects who are still symptomatic (WHO FC II to IV) and have PVR≥ 240 dyn.sec.cm-5 at week 16 will be offered additional treatment by BPA.

Safety follow-up period: After study drug discontinuation, all subjects will enter a Safety follow-up period which ends with safety follow up visit/end of study, 30-35 days after the last intake to the study drug.

All subjects who prematurely and definitively discontinue study drug before Week 42 must have a premature EOT visit as soon as possible but no later than 7 days after the decision of definitive discontinuation of study drug and have a safety follow-up visit as described above.

Post-Treatment Observational Period: Subjects are to remain in the study after premature EOT and safety visit and undergo all study assessments up to Week 42, except subjects discontinuing study drug due to PH-related disease progression who will have a premature EOT visit and Safety follow-up visit and will be withdrawn from the study.

A total of 96 newly diagnosed and treatment-naïve subjects with inoperable CTEPH will be randomly assigned in a 1:1 ratio to receive either macitentan (n=48) or placebo (n=48) combined with standard of care with riociguat.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Male or female ≥18 and ≤ 80 years of age at inclusion.
3. Newly diagnosed and treatment-naïve subjects with CTEPH judged as inoperable due to surgically inaccessible lesions but eligible for balloon pulmonary angioplasty, riociguat and macitentan by multidisciplinary team assessment and fulfilling the following criteria:

   1. Symptomatic pulmonary hypertension (PH) in WHO FC ≥ II.
   2. Confirmation of diagnosis based on 2 of the 3 following methods:

   i. Ventilation-perfusion lung scan ii. Digital subtraction pulmonary angiography (DSA) iii. CT pulmonary angiography (CTPA).
4. Confirmation of inoperability based on CTPA scan and/or DSA.
5. Right-heart catheterization (RHC) in the 12-week period prior to screening visit or during screening period showing the following:

   1. Mean pulmonary artery pressure (mPAP) ≥ 25 mmHg
   2. Pulmonary artery wedge pressure (PAWP) ≤ 15 mmHg or left ventricular end diastolic pressure ≤ 15 mmHg
   3. PVR at rest ≥ 400 dyn.sec.cm-5.
6. Subject anticoagulated (with either vitamin K antagonists or direct oral anticoagulants [e.g., factor IIa inhibitors, factor Xa inhibitors]), or treated with unfractionated heparin or low molecular weight heparin for at least 3 months prior to baseline RHC.
7. 6MWD ≥ 50m
8. Women of childbearing potential must:

   1. Have a negative pre-treatment serum pregnancy test
   2. Agree to use reliable contraception from screening up to 1 month following discontinuation of the last study treatment.

Exclusion Criteria:

1. Previous pulmonary endarterectomy.
2. Previous balloon pulmonary angioplasty.
3. Any PAH-targeted therapy (e.g., any endothelin receptor antagonist (ERA), phosphodiesterase-5 inhibitor (PDE-5i), soluble guanylate cyclase stimulator, prostacyclin, prostacyclin analog, or prostacyclin receptor agonist) at any time prior to inclusion.
4. Ongoing or planned treatment with organic nitrates.
5. Known moderate-to-severe restrictive lung disease (i.e., total lung capacity < 60% of predicted value) or obstructive lung disease (i.e., forced expiratory volume in one second [FEV1] < 60% of predicted, with FEV1 / forced vital capacity < 65%) or known significant chronic lung disease diagnosed by chest imaging (e.g., interstitial lung disease, emphysema).
6. Symptomatic coronary artery disease requiring nitrate use or intervention (e.g., Percutaneous Coronary Intervention, Coronary Artery Bypass Graft) anticipated in the 6-month period after inclusion.
7. Acute myocardial infarction ≤ 12 weeks prior to inclusion.
8. Left heart failure with an ejection fraction less than 40%.
9. Cerebrovascular events (e.g., transient ischemic attack, stroke) ≤ 12 weeks prior to inclusion.
10. History of life-threatening hemoptysis (>100 mL in 24 h) or subjects who have previously undergone bronchial arterial embolization for hemoptysis.
11. Hemoglobin < 100 g/L.
12. Serum aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 3 × upper limit of the normal range.
13. Documented severe hepatic impairment (with or without cirrhosis) according to National Cancer Institute organ dysfunction working group criteria, defined as total bilirubin > 3 × upper limit of the normal range (ULN) accompanied by aspartate aminotransferase (AST) > ULN; and/or Child-Pugh Class C.
14. Severe renal impairment (estimated creatinine clearance ≤ 30 mL/min/1.73 m²).
15. Systolic blood pressure <95mmHg.
16. Treatment with strong cytochrome P450 3A4 (CYP3A4) inducers (e.g., rifabutin, rifampicin, carbamazepine, phenobarbital, phenytoin, St. John's wort) ≤ 28 days prior to inclusion.
17. Treatment with strong multi pathway P-glycoprotein (P-gp)/ breast cancer resistance protein (BCRP) inhibitors (e.g., lopinavir/ritonavir) ≤ 28 days prior to inclusion.
18. Treatment with a strong CYP3A4 inhibitor (e.g., ketoconazole, itraconazole, voriconazole, clarithromycin, telithromycin, nefazodone, ritonavir, and saquinavir) or a moderate dual CYP3A4/CYP2C9 inhibitor (e.g., fluconazole, amiodarone) or co-administration of a combination of moderate CYP3A4 and moderate CYP2C9 inhibitors ≤ 28 days prior to inclusion.
19. Known hypersensitivity to riociguat or macitentan or to any excipient of their formulation.
20. History of severe allergic-like reaction to intravascular administration of iodinated contrast media (including diffuse edema or facial edema with dyspnea, diffuse erythema with hypotension, laryngeal edema with stridor and/or hypoxia, bronchospasm, anaphylactic shock with hypotension and tachycardia).
21. Subject who cannot remain in a supine position for at least 120 min for any reason.
22. Pregnancy, breastfeeding, or intention to become pregnant during the study.
23. Subjects with underlying medical disorders and anticipated life expectancy < 12 months (eg active cancer disease with localized and/or metastasized tumor mass).
24. Alcohol abuse (at investigator discretion)
25. Subject not covered by social security service.
26. Any factor or condition likely to affect protocol compliance of the subject, as judged by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2025-07-03 (Actual); Study Completion 2025-07-03 (Actual)

PRIMARY OUTCOMES:
To compare the effect of an initial dual oral treatment (riociguat, macitentan) vs. standard-of-care initial oral monotherapy (riociguat, placebo) on pulmonary vascular resistance (PVR) prior to BPA. | Week 16
  Pulmonary vascular resistance (PVR) at rest at week 16 expressed as a percentage of the baseline resting PVR.

SECONDARY OUTCOMES:
To compare the effect of an initial dual oral treatment (riociguat, macitentan) vs. standard-of-care initial oral monotherapy (riociguat, placebo) on other clinical measures of pulmonary hypertension prior to BPA | Week 16
  Change from Baseline to Week 16 in 6 Minutes Walk Distance Test
To compare the effect of an initial dual oral treatment (riociguat, macitentan) vs. standard-of-care initial oral monotherapy (riociguat, placebo) on other clinical measures of pulmonary hypertension prior to BPA | Week 16
  Change from Baseline to Week 16 in World Health Organization Functional Classification
To compare the effect of an initial dual oral treatment (riociguat, macitentan) vs. standard-of-care initial oral monotherapy (riociguat, placebo) on other clinical measures of pulmonary hypertension prior to BPA | Week 16
  Change from Baseline to Week 16 in Borg dyspnea score
To compare the effect of an initial dual oral treatment (riociguat, macitentan) vs. standard-of-care initial oral monotherapy (riociguat, placebo) on other clinical measures of pulmonary hypertension prior to BPA | Week 16
  Change from Baseline to Week 16 in NT pro-BNP level
To compare the effect of an initial dual oral treatment (riociguat, macitentan) vs. standard-of-care initial oral monotherapy (riociguat, placebo) on quality of life prior to BPA | Week 16
  Change from Baseline to Week 16 in EuroQol-5D-3Level scale
To compare the effect of an initial dual oral treatment (riociguat, macitentan) vs. standard-of-care initial oral monotherapy (riociguat, placebo) on other clinical measures of pulmonary hypertension after potential BPA | Week 42
  Change from Baseline to Week 42 in 6 Minutes Walk Distance Test
To compare the effect of an initial dual oral treatment (riociguat, macitentan) vs. standard-of-care initial oral monotherapy (riociguat, placebo) on other clinical measures of pulmonary hypertension after potential BPA | Week 42
  Change from Baseline to Week 42 in World Health Organization Functional Classification
To compare the effect of an initial dual oral treatment (riociguat, macitentan) vs. standard-of-care initial oral monotherapy (riociguat, placebo) on other clinical measures of pulmonary hypertension after potential BPA | Week 42
  Change from Baseline to Week 42 in Borg dyspnea score
To compare the effect of an initial dual oral treatment (riociguat, macitentan) vs. standard-of-care initial oral monotherapy (riociguat, placebo) on other clinical measures of pulmonary hypertension after potential BPA | Week 42
  Change from Baseline to Week 42 in NT pro BNP level
To compare the effect of an initial dual oral treatment (riociguat, macitentan) vs. standard-of-care initial oral monotherapy (riociguat, placebo) on quality of life after potential BPA | Week 42
  Change from Baseline to Week 42 in EuroQol-5D-3Level scale
To compare the effect of an initial dual oral treatment (riociguat, macitentan) vs. standard-of-care initial oral monotherapy (riociguat, placebo) on Pulmonary vascular resistance after potential BPA | Week 42
  Change from baseline to week 42 in PVR and percentage of subjects reaching PVR<240 dyn.sec.cm-5 at week 42.
To compare the effect of an initial dual oral treatment (riociguat, macitentan) vs. standard-of-care initial oral monotherapy (riociguat, placebo) on the rate of BPA procedure-related complications | Immediately after intervention
  Frequency and type of BPA procedure-related complications from BPA procedure to end-of-study
To compare the effect of an initial dual oral treatment (riociguat, macitentan) vs. standard-of-care initial oral monotherapy (riociguat, placebo) on the disease progression | Week 42
  Time from randomization to the first PH-related disease progression event up to end-of-study, defined as any of the following :
  Death (all causes), Need for lung transplantation, Hospitalization due to PH, Initiation of parenteral prostanoid therapy due to PH-related disease progression
  , Worsening defined as a post-baseline decrease in 6MWD by ≥ 15 % combined with WHO FC III or IV).
Recording of serious and non serious adverse events/effects, Treatment-emergent adverse events (AEs) and serious adverse events (SAEs), AEs leading to premature discontinuation of study drug | Week 42
Change from baseline in laboratory variable, weight and vital signs o Change from baseline in laboratory variables o Change from baseline in weight and vital signs (arterial blood pressure, heart rate). | Week 42

CONTACTS AND LOCATIONS:
Overall Officials: Xavier JAIS, Dr, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Bicêtre, Le Kremlin-Bicêtre, Île-de-France Region, France